CLINICAL TRIAL: NCT06223711
Title: Durvalumab (MEDI4736) in Combination With Consolidative Radiochemotherapy and Ablative Stereotactic Radiotherapy in Extensive Stage SCLC
Brief Title: Durvalumab With Consolidative Radiochemotherapy and Ablative Stereotactic Radiotherapy in Oligometastatic ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DuCoRa-SCLC
Record Dates: First submitted 2023-12-01; First posted 2024-01-25 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — durvalumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Thoracic Radiochemotherapy concomitant 2 cycles of etoposide/platinum + durvalumab
  Stereotactic radiotherapy of further tumor locations + durvalumab maintenance
  Interventions: Radiation: Thoracic Radiochemotherapy; Drug: durvalumab; Radiation: Stereotactic radiotherapy of further tumor locations; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Thoracic Radiochemotherapy — Radiotherapy to the primary tumor including mediastinal lymph node metastases is delivered in single fractions of 1.8Gy once daily up to a cumulative dose of 63.0Gy by intensity modulated radiation therapy (IMRT) or volumetric modulated arc therapy (VMAT).
Drug: durvalumab — Durvalumab is administered in fixed dose 1500mg in q3w cycles concomitant to chemotherapy and q4w cycles during maintenance treatment
Radiation: Stereotactic radiotherapy of further tumor locations — Stereotactic radiotherapy is delivered to the up to four further tumor locations during durvalumab maintenance therapy and will be performed according to local standards with established dose and fractionation schemes in ablative doses depending on the affected organ system.
Drug: Chemotherapy — Concomitant chemotherapy consists of further two cycles platinum/etoposide q3w (summarized cycle 3-4).

SUMMARY:
Open-label, single-arm, prospective multicenter phase II clinical trial to determine the efficacy of immunotherapy with durvalumab concomitant with radiochemotherapy, followed by durvalumab maintenance therapy in combination with stereotactic radiotherapy in extensive stage SCLC

DETAILED DESCRIPTION:
This is an open-label, prospective, multi-center single-arm phase II trial. Patients with oligometastatic extensive stage SCLC will be enrolled in the trial. In this trial oligometastatic disease is defined as up to five tumor lesions, whereas the primary tumor including mediastinal lymph node metastases counts as one tumor lesion. The primary tumor including lymph node metastases must be suitable for radiochemotherapy and all distant metastases for stereotactic radiotherapy. Patients must have completed systemic therapy with two cycles of platinum/etoposide/durvalumab and have stable disease or partial response according to RECIST 1.1 criteria. After study inclusion, patients receive radiochemotherapy with concomitant durvalumab (MEDI4736). Concomitant chemotherapy consists of further two cycles platinum/etoposide q3w (summarized cycle 3-4). Dosing of chemotherapy is etoposide 90mg/m² body surface area (BSA) day 1-3 in combination with cisplatin 75mg/m² BSA on day 1 or carboplatin area under the curve (AUC) 5 mg/ml per minute on day 1. Split dose of platinum chemotherapy to 2-3 days is an allowed treatment option. Durvalumab is administered in fixed dose 1500mg in q3w cycles concomitant to chemotherapy and q4w cycles during maintenance treatment. Radiotherapy to the primary tumor including mediastinal lymph node metastases is delivered in single fractions of 1.8Gy once daily up to a cumulative dose of 63.0Gy by intensity modulated radiation therapy (IMRT) or volumetric modulated arc therapy (VMAT). In the following, stereotactic radiotherapy is delivered to the up to four further tumor locations during durvalumab maintenance therapy. Sequencing of radiotherapy of the primary tumor and metastases may be changed if radiotherapy of brain, vertebral or other symptomatic metastases is urgently necessary. Stereotactic radiotherapy will be performed according to local standards with established dose and fractionation schemes in ablative doses depending on the affected organ system.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study patients must fulfill all of the following criteria:

1. Histologically confirmed first diagnosis of ES-SCLC according to the Veterans Administration Lung Study Group (VALG) Staging System for SCLC1 (disease extension that cannot be treated within one radiation field).
2. Oligometastatic disease defined as follows:

   * Primary tumor with or without mediastinal or supraclavicular lymph node metastases (counts as one lesion if it can be treated within one radiation field).
   * Up to four distant tumor lesions/metastases that can be treated with stereotactic radiotherapy (stereotactic radiotherapy of lung metastases in addition to radiochemotherapy of primary tumor should previously be discussed with the principal investigator).
   * No cytologically confirmed malignant pleural effusion (in case of suspected malignant pleural effusion in imaging, pleurocentesis for cytological assessment is required).
3. Stable disease (SD) or partial response (PR) according to RECIST 1.1 criteria after previous treatment with two cycles of platinum/etoposide/durvalumab.
4. Adequate lung function defined as forced expiratory volume in the first second (FEV1) ≥1.3 liter in spirometry.
5. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent including European Union Data Privacy Directive obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
6. Age > 18 years at time of study entry.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Body weight >30 kg.
9. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥9.0 g/dL
   * White Blood Cells (WBC) ≥ 3,000 per mm3
   * Platelet count >100,000 per mm3
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
   * Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.
11. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Participation in another clinical study with an investigational product during the last 4 weeks.
2. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Prior systemic anticancer therapy (chemotherapy, immunotherapy, targeted therapy), apart from two cycles of etoposide/platinum + durvalumab (prior chemotherapy/ immunotherapy/ targeted therapy for other malignancy treated with curative intent ≥5 years ago is no exclusion criterion).
4. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous chemo-immunotherapy (2 cycles of platinum/etoposide + durvalumab) with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
5. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
6. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
7. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
8. History of allogenic organ transplantation.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g., colitis or Crohn's disease), diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.). The following are exceptions to this criterion:

   1. Patients with vitiligo or alopecia
   2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   3. Any chronic skin condition that does not require systemic therapy
   4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   5. Patients with celiac disease controlled by diet alone
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active symptomatic infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, QTcF (QT interval on ECG corrected using the Frederica's formula) >470 ms, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
12. History of leptomeningeal carcinomatosis.
13. History of active primary immunodeficiency.
14. Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
15. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings).
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
19. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
20. Prior randomization or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
21. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.
22. Known allergy or hypersensitivity to IP or any excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate | 12 month
  Efficacy of a treatment scheme consisting of thoracic radiotherapy concomitant to platinum/etoposide/durvalumab therapy followed by stereotactic radiotherapy concomitant to durvalumab maintenance to improve the one year PFS rate using investigator assessments according to RECIST 1.1

SECONDARY OUTCOMES:
overall survival (OS) | 12 month
  One-year OS rate

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - University Hospital Augsburg, Radiation Oncology, Augsburg, Bavaria
  - University Hospital Erlangen, Radiation Oncology, Erlangen, Bavaria
  - University Hospital Regensburg, Clinic and Polyclinic for Radiotherapy, Regensburg, Bavaria
  - Kliniken Maria Hilf, Mönchengladbach, North Rhine-Westphalia
  - Saarland University Medical Center and Saarland University Faculty of Medicine, Clinic for Radiotherapy and Radiooncology, Homburg, Saarland